CLINICAL TRIAL: NCT06892821
Title: Prospective Cohort Study of Children Diagnosed with Type 1 Diabetes in Türkiye Between 2018 to 2022
Status: Completed | Type: Observational
Sponsor: Turkish Pediatric Diabetes Working Group (Other)
Responsible Party: Principal Investigator, nursel muratoğlu şahin, Associate Professor, Department of Pediatric Endocrinology, University of Health Sciences, Turkish Pediatric Diabetes Working Group
Other Study IDs: ZTB14/2018
Record Dates: First submitted 2025-03-18; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Type 1 Diabetes Mellitus (T1DM)
Keywords: type 1 diabetes mellitus; children; adolescent
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Achieving glycemic targets with improved T1DM management reduces diabetes complications and the risk of progression. Thus, it is essential to identify the challenges in T1DM management within the country and develop strategies for improvement. In Türkiye, there is limited multicenter data regarding the clinical characteristics of children and adolescents with T1DM during the diagnosis and treatment process. This multicenter prospective cohort study aimed to determine the diagnostic and follow-up characteristics of children and adolescents with T1DM, assess the status of diabetes management in the country.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus can develop in individuals between the ages of 2 months and 18 years.

Exclusion Criteria:

* other types of diabetes mellitus

Ages: 2 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: patients diagnosed with type 1 diabetes mellitus between 01.01.2018 and 31.12.2022 at 42 pediatric diabetes centers across 7 regions of Türkiye
Sampling Method: Probability Sample
Enrollment: 2730 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
HbA1c | Through study completion, HbA1c will be measured during the 1st, 2nd, 3rd, 4th, and 5th years of treatment.
diabetes microvascular complications | through study completion, diabetes microvascular complications will be assessed during the 1st, 2nd, 3rd, 4th, and 5th years of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Ministry of Health Etlik City Hospital, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No